CLINICAL TRIAL: NCT02161107
Title: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled Parallel-Group Study to Assess the Safety and Tolerability of Grass-SPIRE in Subjects With Asthma and Grass-Induced Rhinoconjunctivitis
Brief Title: Study of Grass-SPIRE in Subjects With Grass Allergies and Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG004
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Seasonal Allergic Rhinitis; Asthma
Keywords: Grass; Allergy; rhinoconjunctivitis; rhinitis; asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma; Hypersensitivity; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Grass-SPIRE 1 (Experimental): Grass-SPIRE regimen 1 given 2 weeks apart
  Interventions: Biological: Grass-SPIRE
- Grass-SPIRE 2 (Experimental): Grass-SPIRE regimen 2 given 2 weeks apart
  Interventions: Biological: Grass-SPIRE
- Placebo (Placebo Comparator): Placebo given 2 weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Grass-SPIRE — Intradermal injection
  Arms: Grass-SPIRE 1; Grass-SPIRE 2
Biological: Placebo — Intradermal injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether it is safe to administer Grass-SPIRE to subjects suffering from both grass allergy and asthma

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years.
* Asthma treated by inhaled SABA or inhaled SABA plus low-medium dose ICS in 6 weeks prior to randomisation.
* A reliable history consistent with moderate to severe rhinoconjunctivitis on exposure to grass for at least the previous two grass seasons.
* Positive skin prick test to grass.
* Grass-specific Immunoglobulin E (IgE) ≥ 0.35 kU/L.

Exclusion Criteria:

* History of life-threatening asthma.
* Uncontrolled asthma according to GINA.
* FEV1 of <70 % of predicted, regardless of the cause.
* Administration of adrenaline (epinephrine) is contraindicated (e.g. subjects with acute or chronic symptomatic coronary heart disease).
* History of severe drug allergy or anaphylactic reaction to food.
* A history of any significant disease or disorder (e.g. immune system, pulmonary, cardiovascular, gastrointestinal, liver, renal, neurological, metabolic, malignant, psychiatric, major physical impairment, history of alcohol or drug abuse)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Throughout subjects participation in the study, approximately 15 weeks

SECONDARY OUTCOMES:
Number of subjects with asthma exacerbations as a measure of safety and tolerability | Throughout subjects participation in the study, approximately 15 weeks
Evaluation of change in lung function as a measure of safety and tolerability | Throughout subjects participation in the study, approximately 15 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Kingston General Hospital, Kingston, Ontario
  - Cheema Research Inc, Mississauga, Ontario
  - Inflamax Research, Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Centre de Recherche Appliquée en Allergie de Québec, Québec, Quebec